CLINICAL TRIAL: NCT00004410
Title: Randomized Study of Tauroursodeoxycholic Acid in Prophylactic Therapy of Total Parenteral Nutrition Associated Cholestasis in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13299; CHMC-C-95-9-9; CHMC-C-CRC-473; CHMC-C-FDR001277
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-08

CONDITIONS: Cholestasis
Keywords: cholestasis; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Cholestasis; Gastrointestinal Diseases; Rare Diseases | interventions — ursodoxicoltaurine

INTERVENTIONS:
Drug: tauroursodeoxycholic acid

SUMMARY:
OBJECTIVES: I. Determine whether infants treated with tauroursodeoxycholic acid (TUDCA) have a lower peak direct bilirubin, ALT, AST, glutamyltranspeptidase levels and a reduced duration of cholestasis compared to the nontreatment arm.

II. Determine the significance of lower birth weight and longer duration of total parenteral nutrition (TPN) on increasing risk of TPN associated cholestasis and increasing benefit from TUDCA therapy.

III. Determine whether TUDCA therapy leads to significant reduction in the appearance of biliary tract sludge and/or stone formation in these infants.

IV. Determine whether TUDCA therapy leads to reduced urinary excretion of potentially hepatotoxic bile acids as compared to the untreated arm matched for birth weight and duration of TPN.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by birth weight.

Patients are randomized in pairs by birth weight to receive either a placebo in arm I or tauroursodeoxycholic acid (TUDCA) in arm II. TUDCA is administered by mouth, nasogastric tube, or gastrostomy tube twice daily. After 2 weeks of therapy, a bile sample is obtained via a duodenal tube. An ultrasound examination of the liver and biliary tract is performed after 2 weeks and every 3 weeks thereafter until discontinuation of therapy or until presence of biliary tract sludge is noted on 2 consecutive examinations.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Hospitalized infants who are anticipated to require total parenteral nutrition for greater than 2 weeks and have: Major gastrointestinal anomalies (gastroschisis, ruptured omphalocele) OR Resection (necrotizing enterocolitis, volvulus)
* No evidence of biliary tract abnormalities
* No evidence of other forms of cholestatic liver disease

--Patient Characteristics--

* Renal: No life threatening renal disease
* Cardiovascular: No life threatening cardiovascular disease
* Other: No multiple congenital abnormalities

Max Age: 20 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 1998-06; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: James Heubi, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio